CLINICAL TRIAL: NCT07146100
Title: Prospective, Open-label, Multicenter Long-term Follow-up Study to Evaluate the Durability of Virologic Response in Participants With Chronic Hepatitis B Previously Treated With AHB-137 Injection
Brief Title: Long-term Follow-up Study to Evaluate Participants With Chronic Hepatitis B (CHB) Previously Treated With AHB-137 Injection
Status: Not yet recruiting | Type: Observational
Sponsor: Ausper Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: AB-10-8004
Record Dates: First submitted 2025-08-19; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants who have previously participated in AHB-137 clinical trials

SUMMARY:
This study is a prospective, open-label, multicenter long-term follow-up study to evaluate the durability of virologic response in subjects with chronic hepatitis B previously treated with AHB-137 injection.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent.
* Participants who have previously received at least one dose of AHB-137 and achieved the complete of partial response in the parent study without rescue medication and who maintained response until the End of Study (EoS) visit in their parent study.

Exclusion Criteria:

* Participants who have/or are currently participating in another interventional clinical study since completing their treatment with AHB-137.
* Suspected for cancer at screening or any condition required hospitalization during this study , or any condition which, in the opinion of the investigator or Medical Monitor, contraindicates their participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have previously participated in AHB-137 clinical trials
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-21 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants maintained complete response(defined as HBsAg < 0.05IU/mL and HBV DNA < lower limit of quantification). | Up to 80 weeks

SECONDARY OUTCOMES:
Proportion of participants achieving and maintaining HBsAg<0.05 IU/mL. | Up to 80 weeks
Time to loss of HBsAg reversion. | Up to 80 weeks
Proportion and time of participants meeting certain test indicators after discontinuation of all CHB treatment. | Up to 80 weeks
Serum levels of HBsAg, HBV DNA, HBV RNA, HBcrAg, HBsAb,HBeAb. | Up to 80 weeks
Changes of the five-level five-dimensional health scale (EQ-5D-5L) instrument in participants compared with baseline. | Up to 80 weeks
Percentage of participants with mutations | Up to 80 weeks
Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAE), adverse events, hepatic endpoint events, deathsand clinically significant examination results. | Up to 80 weeks
  Examination including laboratory examination, electrocardiogram (ECG) examination.
Changes of the hepatitis B quality of life (HBQOL) instrument in participants compared with baseline. | Up to 80 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, Principal Investigator — Nanfang Hospital, Southern Medical University; Junqi Niu, Principal Investigator — The First Hospital of Jilin University
Locations (2):
- China (2):
  - AusperBio Investigational Site, Guangzhou, Guangdong
  - AusperBio Investigational Site, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No